CLINICAL TRIAL: NCT01441856
Title: The ORANGE II PLUS - Trial: an International Multicenter Randomized Controlled Trial of Open Versus Laparoscopic Hemihepatectomies.
Brief Title: The ORANGE II PLUS - Trial: Open Versus Laparoscopic Hemihepatectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: University Hospital Southampton NHS Foundation Trust (Other); University Hospital, Ghent (Other); San Raffaele University Hospital, Italy (Other); Derriford Hospital (Other); Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); Queen Elizabeth Hospital NHS Foundation Trust (Other); King's College London (Other); Newcastle-upon-Tyne Hospitals NHS Trust (Other); Oslo University Hospital (Other); General Hospital Groeninge (Other); Jessa Hospital (Other); Universitair Ziekenhuis Brussel (Other); University Hospital, Aachen (Other); Liverpool University Hospitals NHS Foundation Trust (Other Government); Oxford University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NL36215.068.11
Record Dates: First submitted 2011-04-27; First posted 2011-09-28 (Estimated); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Liver Lesions Requiring Hemihepatectomy
Keywords: Open; Laparoscopic; Hemihepatectomy; Hepatectomy; Enhanced Recovery After Surgery; Functional recovery

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: The patient, surgical ward physician and surgical ward nurses are blinded up and until postoperative day 4.
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Open or Laparocopic Left (Active Comparator): Open or Laparoscopic left hemihepatectomy
  Interventions: Procedure: Open or Laparoscopic left hemihepatectomy
- Open or Laparoscopic Right (Active Comparator): Open or Laparoscopic right hemihepatectomy
  Interventions: Procedure: Open or Laparoscopic right hemihepatectomy
- Prospective registry (Active Comparator): Prospective registry of patients that cannot be randomized (both open and laparoscopic left + right hemihepatectomy)
  Interventions: Procedure: Open or Laparoscopic left hemihepatectomy; Procedure: Open or Laparoscopic right hemihepatectomy

INTERVENTIONS:
Procedure: Open or Laparoscopic left hemihepatectomy — Patients in this arm will undergo a left hemihepatectomy within an Enhanced Recovery After Surgery Program.
  Arms: Open or Laparocopic Left; Prospective registry
Procedure: Open or Laparoscopic right hemihepatectomy — Patients in this arm will undergo a right hemihepatectomy within an Enhanced Recovery After Surgery Program.
  Arms: Open or Laparoscopic Right; Prospective registry

SUMMARY:
The added value of the laparoscopic hemihepatectomy compared to the open hemihepatectomy has never been studied in a randomized controlled setting. Therefore, the multicenter international ORANGE II PLUS - trial has been constructed and will provide evidence on the merits of laparoscopic versus open hemihepatectomy in terms of time to functional recovery, hospital length of stay, intraoperative blood loss, operation time, resection margin, time to adjuvant chemotherapy initiation, readmission percentage, (liver-specific) morbidity, quality of life, body image, reasons for delay of discharge after functional recovery, long term incidence of incisional hernias, hospital and societal costs during one year and overall five-year survival.

DETAILED DESCRIPTION:
Liver resection for colorectal metastasis is the only potentially curative therapy and has become the standard of care in appropriately staged patients, offering 5-year survival rates of approximately 35-40%. Also for symptomatic benign lesions and those of uncertain nature or large size, liver resection is a widely accepted treatment. Open hepatectomy (OH) is the current standard of care for the management of primary and secondary malignancies. Although the feasibility of laparoscopic hepatectomy (LH) has been established, only select centres have used this technique as their primary modality.

Laparoscopic liver resection was first reported in 1991. Over the last decade the method has gained wide acceptance for various liver resection procedures. Multiple retrospective case series and reviews comparing open with laparoscopic liver resection indicate that laparoscopic liver resection can be applied safely for both malignant and benign liver lesions. Laparoscopic liver resection has been associated with shorter hospital length of stay, reduced intraoperative blood loss, less postoperative pain, earlier recovery and better quality of life. Initially the left lateral segments of the liver were chosen for anatomic laparoscopic resection with good results. Many liver centres worldwide are currently adopting laparoscopic surgery for resection of anterior segments, but relatively low volumes to operate on, a significant learning curve and lack of evidence restrict the majority of liver surgeons to further adopt and disseminate this technique.

Recently, indications for resectability have been broadened by new (neo)adjuvant chemotherapies and (radio)embolisation techniques. A new impulse for the laparoscopic management of liver lesions came after the first reports of laparoscopic hemihepatectomies. Major hepatic resections can be technically demanding and hold an increased risk for morbidity. It was demonstrated that in expert hands major anatomical laparoscopic liver resections were feasible with good efficacy and safety. Expert liver centers are already performing laparoscopic (extended) hemihepatectomies. Currently, in European centers, a median hospital length of stay of 6.0 to 13.1 and 3.5 to 10.0 days is observed after respectively open and laparoscopic hepatic resection. In expert hands median duration of admission after major hepatic resection varies between 6 - 12.5 for open and 4 - 8.2 for laparoscopic surgery. However, reports are scarce and level 1 evidence on this matter is still to be presented.

Within the framework of optimising postoperative recovery, broader indications for resection and further adoption of laparoscopic liver surgery there is a need for a randomized trial.Regarding postoperative care, enthusiasm has arisen for the Enhanced Recovery After Surgery (ERAS®) program. This multimodal program, derived from Kehlet's 1990's pioneer work in the multimodal surgical care field, involves optimization of several aspects of the perioperative management of patients undergoing major abdominal surgery. In patients undergoing segmental colectomy, the ERAS® -program enabled earlier recovery and consequently shorter hospital length of stay. Furthermore, a reduction of postoperative morbidity in patients undergoing intestinal resection was reported. These results stimulated liver surgeons of the ERAS® group (Maastricht, Edinburgh and Tromsö) to adapt the ERAS®-program to patients undergoing open liver resection. Van Dam et al. found a significantly reduced hospital length of stay after open liver resection when patients were managed within a multimodal ERAS®-program. Besides a reduction of median total hospital length of stay from 8 to 6 days (25%), the data also suggested that a further reduction of stay could be possible as there was a delay between recovery and actual discharge of the patients. Moreover, Stoot et al. showed - retrospectively - a further reduction in length of stay from 7 days to 5 days when patients were operated laparoscopically and managed within an ERAS®-program. In this study there was also a delay between recovery and actual discharge of the patients. Earlier, Maessen et al. reported a median delay to discharge of 2 days after patients had functionally recovered from colonic surgery managed within an ERAS®-program. This delay is often linked to social problems, problems in homecare support or logistic problems.

The added value of the laparoscopic hemihepatectomy compared to the open hemihepatectomy has never been studied in a randomized controlled setting. Therefore, the multicenter international ORANGE II PLUS - trial has been constructed and will provide evidence on the merits of laparoscopic versus open hemihepatectomy.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring open or laparoscopic left / right hemihepatectomy, with or without the need for one additional hepatic wedge resection or metastasectomy, for accepted indications.
* Able to understand the nature of the study and what will be required of them.
* Men and non-pregnant, non-lactating women age 18 years and older.
* BMI between 18-35.
* Patients with ASA I-II-III.

Exclusion Criteria:

* Inability to give written informed consent.
* Patients undergoing liver resection other than left or right hemihepatectomy, with or without the need for one additional hepatic wedge resection or metastasectomy.
* Patients with hepatic lesion(s), that are located with insufficient margin from vascular or biliary structures to be operated laparoscopically.
* Patients with ASA IV-V.
* Repeat hepatectomy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2013-10-01 (Actual); Primary Completion 2019-12-04 (Actual); Study Completion 2023-12-04 (Actual)

PRIMARY OUTCOMES:
Time to functional recovery | expected average of 4-10 days
  Time until a patient is functionally recovered

SECONDARY OUTCOMES:
Length of hospital stay | 30 days
  Total length of hospital stay
Readmission percentage | 1 year
  Total percentage of patients being readmitted
Total morbidity | 1 year
  Total morbidity during one year
Composite endpoint of liver specific morbidity | 1 year
  Composite endpoint of liver specific morbidity(intra-abdominal bleeding, intra-abdominal abcess, ascites, postresectional liver failure, intra-operative mortality, bile leakage)
Long term incidence of incisional hernia | 1 year
  Incidence of incisional hernia after 1 year
Quality of life: QLQ-C30 + LM 21 | 1 year
  Quality of life assessment (QLQ-C30 + LM 21) during one year
Body image and cosmesis | 1 year
  Influence of intervention on body image and cosmesis during one year
Reasons for delay in discharge after functional recovery | 1 year
Intraoperative blood loss | During procedure
Intraoperative time | Surgical time from incision to closure
Resection margin | During pathology assessment
Time to adjuvant chemotherapy initiation | 1 year
Disease-free survival | 1 year
Hospital and societal costs | 1 year
Overall survival | 1 year and 5 years

CONTACTS AND LOCATIONS:
Overall Officials: R.M. van Dam, MD PhD, Principal Investigator — Maastricht University Medical Center
Locations (16):
- Belgium (4):
  - Erasmus Hospital, Brussels
  - Ghent University Hospital, Ghent
  - Jessa Hospital, Hasselt
  - General Hospital Groeninge, Kortrijk
- University Hospital Aachen, Aachen, Germany
- San Raffaele Hospital, Milan, Italy
- Netherlands (2):
  - Academic Medical Center, Amsterdam
  - Maastricht University Medical Center+, Maastricht
- University Hospital Oslo, Oslo, Norway
- United Kingdom (7):
  - Aintree University Hospital, Aintree
  - Queen Elizabeth Hospital, Birmingham
  - King's College Hospital, London
  - Freeman Hospital, Newcastle
  - Oxford University Hospitals, Oxford
  - Derriford Hospital, Plymouth
  - University Hospital Southampton, Southampton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Olij B, Pilz da Cunha G, Kimman M, Ratti F, Abu Hilal M, Troisi RI, Sutcliffe RP, Besselink MG, Aroori S, Menon KV, Edwin B, D'Hondt M, Lucidi V, Ulmer TF, Diaz-Nieto R, Soonawalla Z, White S, Sergeant G, Coolsen MME, Kuemmerli C, Scuderi V, Berrevoet F, Vanlander A, Marudanayagam R, Tanis PJ, Dewulf MJL, Fichtinger RS, Eminton ZB, Neumann UP, Brandts L, Pugh SA, Fretland AA, Primrose JN, van Dam RM; ORANGE II PLUS Collaborative. Healthcare Utilization, Costs, and Cost-Effectiveness of Patients Undergoing Laparoscopic and Open Hemihepatectomy: A Secondary Analysis of the ORANGE II PLUS Randomized Controlled, Phase 3, Superiority Trial. Ann Surg Oncol. 2025 Dec 12. doi: 10.1245/s10434-025-18779-4. Online ahead of print. PMID 41385067
- [Derived] Olij B, Fichtinger RS, Aldrighetti LA, Abu Hilal M, Troisi RI, Sutcliffe RP, Besselink MG, Aroori S, Menon KV, Edwin B, D'Hondt M, Lucidi V, Ulmer TF, Diaz-Nieto R, Soonawalla Z, White S, Sergeant G, Ratti F, Kuemmerli C, Scuderi V, Berrevoet F, Vanlander A, Marudanayagam R, Tanis PJ, Dewulf MJL, Eminton ZB, Neumann UP, Brandts L, Pugh SA, Fretland AA, Kimman ML, Primrose JN, van Dam RM; ORANGE II PLUS Collaborative. Health-related quality of life in patients undergoing laparoscopic versus open hemihepatectomy: a secondary analysis of the ORANGE II PLUS randomised controlled, phase 3, superiority trial. Lancet Reg Health Eur. 2025 May 19;54:101311. doi: 10.1016/j.lanepe.2025.101311. eCollection 2025 Jul. PMID 40491830
- [Derived] Fichtinger RS, Aldrighetti LA, Abu Hilal M, Troisi RI, Sutcliffe RP, Besselink MG, Aroori S, Menon KV, Edwin B, D'Hondt M, Lucidi V, Ulmer TF, Diaz-Nieto R, Soonawalla Z, White S, Sergeant G, Olij B, Ratti F, Kuemmerli C, Scuderi V, Berrevoet F, Vanlander A, Marudanayagam R, Tanis P, Dewulf MJL, Dejong CHC, Eminton Z, Kimman ML, Brandts L, Neumann UP, Fretland AA, Pugh SA, van Breukelen GJP, Primrose JN, van Dam RM; ORANGE II PLUS Collaborative. Laparoscopic Versus Open Hemihepatectomy: The ORANGE II PLUS Multicenter Randomized Controlled Trial. J Clin Oncol. 2024 May 20;42(15):1799-1809. doi: 10.1200/JCO.23.01019. Epub 2024 Apr 19. PMID 38640453